CLINICAL TRIAL: NCT00762970
Title: Controlling Myopia Progression With Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-1561AB
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Lens 1 (Experimental): Investigational soft contact lenses worn daily.
  Interventions: Device: Test Lens 1
- Test Lens 2 (Experimental): Investigational soft contact lenses worn daily.
  Interventions: Device: Test Lens 2
- Control lens (Active Comparator): Spectacle lenses worn daily.
  Interventions: Device: Control Lens

INTERVENTIONS:
Device: Test Lens 1 — Investigational soft contact lens with asperic optical design to control myopia progression.
  Arms: Test Lens 1
Device: Test Lens 2 — Investigational soft contact lens with asperic optical design to control myopia progression.
  Arms: Test Lens 2
Device: Control Lens — Spectacle Lenses.
  Arms: Control lens

SUMMARY:
This study is to investigate whether novel soft contact lens optical designs can slow myopia progression.

DETAILED DESCRIPTION:
The study will be a prospective, randomized, single blind, bilateral dispensing study

ELIGIBILITY:
Inclusion Criteria:

1. Myopic subjects between 8 and 12 years of age.
2. The subject best sphere contact lens correction must lie between -0.75D (best of the two eyes) and -5.00D (worst of the two eyes)
3. Astigmatism must be less than or equal to 1.00D
4. 1.00D or less difference in spherical equivalent between the two eyes
5. The subject must have a best-corrected visual acuity of 0.8+2 (20/25+2) and spherical equivalent refraction visual acuity of 0.820/25) or better in both eyes
6. The subject must have at least 8D of accommodation
7. The subject and subject's parent or legal guardian must read and sign the STAEMENT OF INFORMED CONSENT
8. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

1. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
2. Systemic disease or autoimmune disease or use of medication (e.g. antihistamine), which may interfere with lens wear.
3. Clinically significant (grade 3 or 4)corneal edema, corneal vascularization, corneal staining, or any other abnormality of the cornea, which may contraindicate contact lens wear.
4. Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection that might interfere with contact lens wear.
5. Any ocular infection.
6. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
7. Any infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g. HIV)
8. Diabetes
9. Anisometropia of greater than 1.00D
10. Astigmatism of greater than 1.00D in either eye
11. Eye injury or surgery within eight weeks immediately prior to enrollment for this study.
12. Pervious refractive surgery, rigi contact lens wear, orthokeratology, keratconus or other corneal irregularity in either eye.
13. Strabismus in either eye
14. Pupil orr lid abnormality or infection in either eye
15. Central corneal scar in either eye
16. Aphakia in either eye
17. Contraindications to contact lens wear such as dry eye or history of prior unsuccessful contact lens wear.
18. History of participation in prior clinical trials aimed to control myopia progression
19. Surgically altered eyes, ocular infection of any type, ocular inflammation
20. Subject has anterior chamber angle grade 2 or narrower

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2010-02-01 (Actual); Study Completion 2010-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Cheng, MD, PhD, Principal Investigator — Principal Clinical Scientist
Locations (1):
- The Tianjin Eye Hospital, Tianjin, China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of those 150 screened subjects, 3 were not eligible to participate in the study and 10 were not randomized to the study lens groups. 115 subjects completed all study visits without a major protocol deviation.
Groups:
- Control Lens: Control spectacle lenses worn daily.
Period: Overall Study
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens
Started | 46 | 44 | 47
Completed | 34 | 35 | 46
Not Completed | 12 | 9 | 1
Not completed — Withdrawal by Subject | 7 | 4 | 0
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Difficulty of handling lens | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on all subjects who randomized in the study.
Groups:
- Test Lens 1; Test Lens 2: Investigational soft contact lens worn daily.
- Total: Total of all reporting groups
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens | Total
Number analyzed (Participants) | 46 | 44 | 47 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 44 | 47 | 137
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (1.1) | 9.8 (1.2) | 9.7 (1.2) | 9.8 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 26 | 78
  Male | 16 | 22 | 21 | 59
Region of Enrollment [Count of Participants; unit: Participants]
  China: Ch | 46 | 44 | 47 | 137

OUTCOME MEASURES:

1. Primary Outcome: Spherical Equivalent Refraction
Description: Spherical equivalent refraction was computed from the sphero-cylindrical refraction measured with an open-field auto refractor (WAM-5500) and descriptively summarized for each follow-up. Higher spherical refraction indicates progression in Myopia.
Time Frame: Baseline and every 6 months post-baseline for 2 years
Population: Analysis was conducted on all randomized subjects who have at least one data point.
Measure: Mean (Standard Deviation); unit: diopter (D)
Units Other Than Participants: eyes
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens
Number analyzed (Participants) | 35 | 37 | 46
Number analyzed (eyes) | 70 | 74 | 92
diopter (D)
  Change from baseline 6 months: number analyzed (eyes) | 68 | 74 | 92
  Change from baseline 6 months | -0.326 (0.6678) | -0.460 (0.3938) | -0.430 (0.3942)
  Change from baseline 12 months: number analyzed (eyes) | 70 | 72 | 90
  Change from baseline 12 months | -0.898 (0.4695) | -0.859 (0.4955) | -0.905 (0.5918)
  Change from baseline 18 months: number analyzed (eyes) | 70 | 72 | 88
  Change from baseline 18 months | -1.222 (0.8501) | -1.185 (0.6550) | -1.336 (0.7361)
  Change from baseline 24 months: number analyzed (eyes) | 48 | 52 | 68
  Change from baseline 24 months | -1.506 (0.9346) | -1.376 (0.5891) | -1.809 (0.9485)

2. Primary Outcome: Axial Length (Axial Elongation)
Description: Axial length was measured with the IOLMaster at baseline and every 6 months post-baseline for 2 years. Axial length was descriptively summarized for each follow-up.
Time Frame: Baseline and every 6 months post-baseline for 2 years
Population: Analysis was conducted on all randomized subjects who have at least one data point.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Units Other Than Participants: eyes
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens
Number analyzed (Participants) | 35 | 37 | 46
Number analyzed (eyes) | 70 | 74 | 92
millimeter (mm)
  Change from baseline 6 months: number analyzed (eyes) | 68 | 74 | 92
  Change from baseline 6 months | 0.214 (0.1020) | 0.198 (0.1128) | 0.263 (0.1766)
  Change from baseline 12 months: number analyzed (eyes) | 70 | 72 | 90
  Change from baseline 12 months | 0.401 (0.1816) | 0.382 (0.1974) | 0.458 (0.2323)
  Change from baseline 18 months: number analyzed (eyes) | 70 | 72 | 88
  Change from baseline 18 months | 0.564 (0.2371) | 0.522 (0.2643) | 0.622 (0.2805)
  Change from baseline 24 months: number analyzed (eyes) | 48 | 52 | 68
  Change from baseline 24 months | 0.660 (0.2355) | 0.529 (0.2378) | 0.749 (0.3203)

ADVERSE EVENTS:
Arm/Group | Test Lens 1 | Test Lens 2 | Control Lens
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/44 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes